CLINICAL TRIAL: NCT01725100
Title: An Open-label, Randomized, 2-treatment, 2-period, 2-way Crossover, Single-dose Study to Determine the Relative Bioavailability of the MEK Inhibitor, Trametinib, in Subjects With Solid Tumor Malignancies
Brief Title: A Study to Determine the Relative Bioavailability of the MEK Inhibitor, Trametinib, in Subjects With Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 114656
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: GSK1120212; DMSO content; pharmacokinetics; solid tumors; MEK inhibitor; dissolution; trametinib; relative bioavailability
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A: GSK1120212B (Standard DMSO content) (Experimental): Subjects will receive Treatment A in Period 1 or 2 as single oral dose on Day 1 of Period 1 or 2 in fasting condition with water.
  Interventions: Drug: GSK1120212B (Standard DMSO content)
- Treatment B: GSK1120212B (Lower DMSO content) (Experimental): Subjects will receive Treatment B in Period 1 or 2 as single oral dose on Day 1 of Period 1 or 2 in fasting condition with water.
  Interventions: Drug: GSK1120212B (Lower DMSO content)

INTERVENTIONS:
Drug: GSK1120212B (Standard DMSO content) — Each tablet contains GSK1120212B equivalent to 2 mg of GSK1120212 as drug substance. The coated tablets have a standard DMSO content of theoretical 11.3%.
  Arms: Treatment A: GSK1120212B (Standard DMSO content)
Drug: GSK1120212B (Lower DMSO content) — Each tablet contains GSK1120212B equivalent to 2 mg of GSK1120212 as drug substance. The coated tablets have a lower DMSO content approximately 9.5%.
  Arms: Treatment B: GSK1120212B (Lower DMSO content)

SUMMARY:
This is an open-label, randomized, single-dose, 2-treatment, 2-period, 2-way crossover study with incomplete wash-out in subjects with solid tumors to determine the relative bioavailability of test formulation with lower dimethyl sulfoxide (DMSO) content as compared with standard reference formulation trametinib.

Approximately 18 subjects will be randomized to receive either a single dose of Treatment A (standard target DMSO content [theoretical 11.3%] formulation of GSK1120212B) or a single dose of Treatment B (lower DMSO Content [approximately 9.5%] formulation of GSK1120212B) followed by a 7 day incomplete wash-out period, then a single dose of the other treatment.

Administration of the dose under fasted conditions in Periods 1 and 2 will be only on Day 1 followed by 7 days of serial blood sampling for PK analysis of plasma trametinib. Safety assessments, including assessment of AEs, clinical laboratory (hematology and clinical chemistry) and vital signs, will be made throughout the study.

After a subject completes the study, he or she may be eligible to enter study MEK114375, an open-label rollover study of trametinib (no wash-out period or follow-up visit required) and continue receiving trametinib. For those subjects who wish to discontinue or complete the current study and choose not enter the rollover study, a follow-up visit should be performed within 21 days after receiving the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has provided signed, written informed consent.
* Male or female, age >=18 years of age at the time of signing the informed consent form.
* Has histologically or cytologically confirmed diagnosis of a solid tumor malignancy that is not responsive to standard therapy (ies) or for which there is no approved therapy.
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal (GI) abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* All prior treatment-related toxicities must be National Cancer Institute - Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 4.0 <=Grade 1 (except alopecia) at the time of enrollment.
* Has adequate baseline organ function as defined: ANC >=1.2×10^9/liter (L), hemoglobin>=9 gram (g)/deciliter (dL), Platelets>=75×10^9/L, partial thromboplastin time (PTT), prothrombin time (PT) and International normalization ratio (INR) <=1.5 times upper limit of normal (ULN), albumin >=2.5 g/dL, total bilirubin <=1.5 times ULN alanine aminotransferase (ALT) <=2.5 times ULN, Creatinine or calculated creatinine clearance >=50 milliliter (mL)/minute (min) and left ventricular ejection fraction (LVEF)>=lower limit of normal (LLN) by echocardiogram (ECHO) or multigated acquisition scan (MUGA).
* Women of childbearing potential must have a negative serum pregnancy test within 14 days of first dose of study treatment and agree to use effective contraception, during the study and for 4 months following the last dose of study treatment.

Exclusion Criteria:

* Prior exposure to a mitogen-activated extracellular signal-regulated kinase (MEK) inhibitor.
* Anti-cancer therapy (e.g., chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy, or major surgery) within 21 days prior to randomization; chemotherapy regimens without delayed toxicity within 14 days prior to randomization.
* Female Subjects: Lactating or actively breastfeeding.
* Has participated in a clinical trial and received investigational drug within 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (IP), whichever is longer, prior to randomization in this study.
* Has participated in a study that resulted in or made a donation of blood or blood products in excess of 500 mL within 56 days of the first dose of study treatment.
* History or presence of hepatic insufficiency (excluding metastatic hepatic carcinoma).
* History of interstitial lung disease or pneumonitis.
* Known Human Immunodeficiency Virus, Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection
* Subjects with laboratory evidence of cleared HBV and HCV infection will be permitted.
* Has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study treatment, or excipients, or to DMSO.
* Currently using a prohibited medication or requires the use of any of the prohibited medications during the study. Use of anticoagulants such as warfarin is permitted provided INR must be monitored in accordance with local institutional practice.
* Has a history of another malignancy. Subjects who have been disease-free for 3 years or subjects with a history of a completely resected non-melanoma skin cancer and/or subjects with indolent second malignancies are eligible.
* Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
* Has a history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR).
* Symptomatic or untreated leptomeningeal or brain metastases, or spinal cord compression.
* Left ventricular ejection fraction (LVEF), as measured by ECHO or MUGA scan, below the institutional LLN, or if a LLN does not exist at an institution, <50%.
* QT interval corrected for heart rate using the Bazett formula (QTcB) >=480 millisecond (msec).
* History or current evidence of cardiovascular risk including any of the following: current clinically significant uncontrolled arrhythmias, acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization, current >= Class II congestive heart failure as defined by New York Heart Association (NYHA), treatment-refractory hypertension defined as a blood pressure of systolic blood pressure (SBP) >140 millimeters of mercury (mmHg) and/or diastolic blood pressure (DBP) >90 mmHg which cannot be controlled by anti-hypertensive therapy, has an intra-cardiac defibrillator or permanent pacemaker and known cardiac metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-02-05 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2015-01-30 (Actual)

PRIMARY OUTCOMES:
Corrected Cmax of GSK1120212B | Period 1 and 2: Day 1 pre-dose within 15 minutes (mins) of planned study treatment administration (serves as the 168-hour [hr] sample for Period 1), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 10 hrs post-dose; Days 2 to 7: post dose at 24 hrs (Day 2), 48 hrs (
  Pharmacokinetic data will include corrected maximum plasma concentration (Cmax) of GSK1120212B. Comparison of Cmax will enable to determine the relative bioavailability of the test formulation with lower DMSO content (Treatment B) and the standard reference formulation (Treatment A). Period 2 PK parameters will be corrected for residual concentrations from Period 1 (based on individual estimates of t1/2) to remove the carry-over effect.
Corrected AUC(0-t) and AUC(0-inf) of GSK1120212B | Period 1 and 2: Day 1 pre-dose within 15 mins of planned study treatment administration (serves as the 168-hr sample for Period 1), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 10 hrs post-dose; Days 2 to 7: post dose at 24 hrs (Day 2), 48 hrs (Day 3), 72 hrs (
  Pharmacokinetic data will include corrected area under the time-concentration curve from time zero (pre-dose) to last time of quantifiable concentration (AUC(0-t)) and AUC from zero to infinity (AUC(0-inf)) of GSK1120212B. Period 2 PK parameters will be corrected for residual concentrations from Period 1 (based on individual estimates of t1/2) to remove the carry-over effect.
Corrected tmax of GSK1120212B | Period 1 and 2: Day 1 pre-dose within 15 mins of planned study treatment administration (serves as the 168-hr sample for Period 1), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 10 hrs post-dose; Days 2 to 7: post dose at 24 hrs (Day 2), 48 hrs (Day 3), 72 hrs (
  Pharmacokinetic data will include corrected time of occurrence of Cmax (tmax) of GSK1120212B. Period 2 PK parameters will be corrected for residual concentrations from Period 1 (based on individual estimates of t1/2) to remove the carry-over effect.

SECONDARY OUTCOMES:
Uncorrected Cmax of GSK1120212B | For Period 1 and 2 on Day 1: pre-dose within 15 mins of planned study treatment administration (serves as the 168-hr sample for Period 1), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 10 hrs post-dose; Days 2 to 7: post dose at 24 hrs (Day 2), 48 hrs (Day 3), 72
  Pharmacokinetic data will include uncorrected Cmax of GSK1120212B.
Uncorrected AUC(0-t), AUC(0-inf) and AUC(0-24) of GSK1120212B | For Period 1 and 2 on Day 1: pre-dose within 15 mins of planned study treatment administration (serves as the 168-hr sample for Period 1), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 10 hrs post-dose; Days 2 to 7: post dose at 24 hrs (Day 2), 48 hrs (Day 3), 72
  Pharmacokinetic data will include uncorrected AUC(0-t), AUC(0-inf) and AUC from zero to 24 hrs AUC(0-24) of GSK1120212B.
Pre-dose concentration (C0) of GSK1120212B | Period 2: Day 1 pre-dose within 15 minutes (mins) of planned study treatment administration (serves as the 168-hour [hr] sample for Period 1.
  Pharmacokinetic data will include uncorrected C0 of GSK1120212B in Period 2
Elimination half life (t½) of GSK1120212B | Period 1 and 2: Day 1 pre-dose within 15 mins of planned study treatment administration (serves as the 168-hr sample for Period 1), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 10 hrs post-dose; Days 2 to 7: post dose at 24 hrs (Day 2), 48 hrs (Day 3), 72 hrs (
  Pharmacokinetic data will include t1/2 of GSK1120212B.
Safety of GSK1120212B as assessed by changes in vital signs measurements | Through Day 36.
  Safety data will include measurements of vital signs (blood pressure, pulse rate and temperature) at Baseline and end of the study.
Safety of GSK1120212B as assessed by changes in clinical laboratory tests | Through Day 36.
  Safety data will include assessments of clinical laboratory tests (hematology, clinical chemistry, coagulation and at Baseline and end of the study.
Safety of GSK1120212B as assessed by number of subjects with adverse events (AE)s | Through Day 36
  Safety data will include recording of number of subjects with AEs.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Goodyear, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Nashville, Tennessee

REFERENCES:
- See also: Results for study 114656 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114656?search=study&search_terms=114656#rs